CLINICAL TRIAL: NCT06054048
Title: Open Video System in Medicine (oVID) - Use Case Palliative Care
Brief Title: Open Video System in Medicine (oVID)
Acronym: oVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Palliativnetz Muenster gGmbH (Unknown); CompuGroup Medical (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EFRE-0801384
Record Dates: First submitted 2023-07-28; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-07

CONDITIONS: Cancer; Chronic Heart Failure; Chronic Obstructive Pulmonary Disease; Palliative Care
MeSH Terms: conditions — Neoplasms; Pulmonary Disease, Chronic Obstructive | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: Randomized controlled non-inferiority trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine (Active Comparator): Those patients who received specialized outpatient palliative care plus telemedicine.
  Interventions: Other: Telemedicine
- No telemedicine (Standard of Care) (No Intervention): Those patients who received standard specialized outpatient palliative care only.

INTERVENTIONS:
Other: Telemedicine — Web Real-Time Communication (WebRTC), which enables a peer-to-peer connectivity. Communication platform for all TCs was the software "CompuGroup Medical Electronic Visit" (CGM ELVI), which provides end-to-end encrypted video conferencing between physicians and their patients.
  Arms: Telemedicine

SUMMARY:
Currently, there are no telemedical visits between patients and/or their relatives and a palliative physician for the evaluation of symptom and progress monitoring. This is done during visits of the patient by the coordinators and palliative physicians of the palliative network/PKD Münster (PKD = Palliative Care Consultation Service) and/or the general practitioners. Upon enrollment in the Palliative Network/PKD Münster, patients receive a 24-hour emergency telephone number. This is staffed by a caregiver who coordinates the deployment of other caregivers / palliative care physicians according to the information provided by the patient / family members. If patients are randomized to the "telemedicine" group, they have the option of using ELVI (ELVI = electronic visit) in addition to conventional care, and thus the possibility of televisits with physicians or nurses. In this case, they receive access data for ELVI, i.e., an access code for a virtual waiting room. In addition, patients will be given questionnaires at discharge to be completed on the day of discharge and on days 7, and 14.

The primary objective of this randomized trial is to demonstrate that telemedically managed patients are not relevantly inferior to conventionally managed patients in terms of change in Integrated Palliative care Outcome Scale (IPOS) from the day of discharge (non-inferiority question), although the possibility of televisiting may result in less frequent physician visits to the patient's home.

DETAILED DESCRIPTION:
Purpose

The increasing specialization of medicine and the growing shortage of medical professionals, especially in rural areas, call for constant networking of clinical facilities. This networking is driven not least by the medical societies. For example, networks have been established throughout Germany in the care of severely injured patients, in neurology, palliative medicine, intensive care medicine, infectious diseases, cardiology and other specialist disciplines. All of these networks aim to improve the joint care of the respective patients, even across sector boundaries.

Moreover, demographic change has been inexorably causing society to age for years. A steadily growing proportion of the population is at an age when the demand for medical treatment is increasing. At the same time, there is a shortage of qualified medical personnel. By 2030, there will be a shortage of up to 106,000 physicians and 575,000 nurses. A double-digit share of all medical positions will probably not be filled. This development is felt with particular intensity in rural areas. Here, the average age of the population and thus the need for medical services, as well as the shortage of doctors and nurses, are even higher than the national average.

In the course of digitization, a wide range of opportunities are opening up that will enable greater efficiency in the treatment of many patients, especially in rural areas. However, the individual networks use heterogeneous, technical systems and standards to a varying extent for this purpose. While the exchange of image data (e.g., X-ray, CT, and MRI examinations) between individual institutions has already become standard in some regions of Germany (e.g., West German Teleradiology Network), there is no communication system that is accessible everywhere and can be used across disciplines, that can be used by every network, that offers the necessary functions, and that can also be adapted to the needs of the respective network. A connection of many different systems is made difficult by high interface, integration and process costs, and in some cases virtually impossible. A system that enables cross-clinic, interdisciplinary communication is not comprehensively available at the present time.

The question of palliative care is becoming increasingly important both in hospitals and in the outpatient setting. Recent studies have shown that palliative care can not only improve the quality of life, but also significantly improve the outcome of treatment and thus prolong survival. Patients with incurable, advanced diseases die more often in hospital than - as often desired - in the home environment. However, both the shortage of physicians and increasing urbanization make it difficult to realize this area-wide provision of palliative care, especially in rural areas. "Communication and shared decision making" and "trust and confidence in treatment partners" are the most important factors for quality end-of-life care. For patients at the end of life, a visit to a (specialist) physician and the associated transport can be a major, energy-sapping and emotional effort. By bringing together various disciplines in one place, as is the case at University Hospital Muenster, and by using telemedical rounds, it may be possible to protect resources on the patient side as well.

Currently, there are no telemedical visits between patients and/or their relatives and a palliative physician for the evaluation of symptom and progress monitoring. This is done during visits of the patient by the coordinators and palliative physicians of the palliative network/PKD Münster and/or the general practitioners. Upon enrollment in the Palliative Network/PKD Münster, patients receive a 24-hour emergency telephone number. This is staffed by a caregiver who coordinates the deployment of other caregivers / palliative care physicians according to the information provided by the patient / family members. If patients are randomized to the "telemedicine" group, they have the option of using ELVI in addition to conventional care, and thus the possibility of televisits with physicians or nurses. In this case, they receive access data for ELVI, i.e., an access code for a virtual waiting room. In addition, patients will be given questionnaires at discharge to be completed on the day of discharge and on days 7, and 14.

The primary objective of this randomized trial is to demonstrate that telemedically managed patients are not relevantly inferior to conventionally managed patients in terms of change in IPOS from the day of discharge (non-inferiority question), although the possibility of televisiting may result in less frequent physician visits to the patient's home.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indications to receive specialized palliative care for advanced malignant and non-malignant diseases
* Minimum age 18 years
* Signed informed consent
* Inpatient care in a normal ward or the palliative care unit at University Hospital Muenster
* Planned discharge to home environment
* Consent to participate in randomized study
* Residence in the area of responsibility of the palliative care network/PKD Münster and consent to the Connection to the palliative care network/PKD Münster
* At least one cell phone (or comparable device with camera and microphone) with wireless network connection or long data evolution (LTE) flat rate
* Basic willingness to use new media
* Disease phase "stable" / "unstable" / "deteriorating" (patients who are in the dying phase are not included in the randomized part of the study, as they will in all likelihood not be discharged home).

Exclusion Criteria:

* Pregnant or breastfeeding patients
* minors
* Language difficulties (lack of German language skills), if these cannot be compensated by family members or interpreters can be compensated
* Dependency or employment relationship to the project management or the including physician
* Persons who have been placed in an institution by court or official order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Symptom Control | 7 days
  Change in the Integrated Palliative Care Outcome Scale (IPOS) over the first seven days after transfer (analyzed for the randomized part of the trial in a non-inferiority analysis). The total scores using IPOS can range between 0 and 68 points. The higher the score, the more severe are the patient's symptoms. IPOS was evaluated using a paper questionnaire. seven days after transfer (analyzed for the randomized part of the trial in a non-inferiority analysis).

SECONDARY OUTCOMES:
Reason for request | up to two weeks
  What were the reasons for requesting the telemedicine rounds?
resulting interventions | up to two weeks
  What actions resulted from the telemedical consultations (e.g., changes in medications, hospitalizations)?
avoidance of home visits | up to two weeks
  How many specialized outpatient palliative care home visits were avoided as a result of telemedical consultations?
number of telephone and visit contacts | up to two weeks
  How many telephone and telemedical consultations have taken place?
sense of safety of patients and professional users | 7 and 14 days
  How was the sense of security among patients and health care workers? (6-point Likert scale (values: 1 (minimum) to 6 (maximum)), lower values mean higher sense of security)

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Lenz, MD, Principal Investigator — University Hospital Muenster
Locations (1):
- University Hospital Muenster, Münster, Germany

REFERENCES:
- [Derived] Bernhardt F, Buckmann A, Kruger J, Bauer B, Hofmeister U, Juhra C, Eveslage M, Fischhuber K, Storck M, Brix TJ, Lenz P. Telemedicine Plus Standard Care Versus Standard Care Only in Specialized Outpatient Palliative Care: A Randomized Controlled Noninferiority Trial. Telemed J E Health. 2024 May;30(5):1459-1469. doi: 10.1089/tmj.2023.0621. Epub 2024 Jan 31. PMID 38294865